CLINICAL TRIAL: NCT05421559
Title: Transection of Sternothyroid Muscle Increases the Rate of Exposure of the External Branch of the Superior Laryngeal Nerve During Thyroidectomy
Brief Title: Transection of Sternothyroid Muscle Increases the Rate of Exposure of the External Laryngeal Nerve During Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Aouf (Other)
Responsible Party: Sponsor-Investigator, Ahmed Aouf, Dr, assistant lecturer of General Surgery, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MKSU50-6-9
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Thyroid; Surgery; Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional approach of thyroidectomy (Active Comparator): conventional method of thyroidectomy with ST muscle retraction
  Interventions: Procedure: thyroidectomy
- transection approach of thyroidectomy (Active Comparator): method of thyroidectomy with ST muscle transection
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — removal of the diseased thyroid gland by conventional method vs transection method of sternothryroid muscle

SUMMARY:
The sternothyroid (ST) muscle is closely adherent to the thyroid gland with oblique insertion into the thyroid cartilage. EBSLN passes through the sternothyroid laryngeal triangle with a parallel course deep to the ST muscle.

This study evaluates the transection of the sternothyroid muscle as a key step during thyroidectomy to increase the rate of exposure and visual identification of EBSLN compared to ST muscle retraction as a traditional technique.

DETAILED DESCRIPTION:
The study was conducted on patients eligible for total thyroidectomy, which meets the standard of the ATA Thyroid Guidelines. Preoperative biochemical thyroid function tests and neck ultrasound with FNAC of suspicious nodules confirmed the clinical diagnosis. Patients who had previously undergone neck surgery or irradiation or were preoperatively diagnosed with a vocal cord movement disorder, a vocal cord benign lesion, or speech disorders were excluded from the study. A random number was used to determine the patient group allocation.

Data about patients were gathered via history, examinations, and investigations. The patients were randomized (computer-generated) with the use of an opaque-sealed envelope into two groups; group A: conventional method of thyroidectomy with ST muscle retraction, group B: transection of ST muscle.

The study's primary endpoint was the identification rate of the EBSLN in both techniques. The secondary endpoints included: a comparison of operative time in both techniques as well as anatomical variability of the EBSLN according to Cernea classification, rate of injury of EBSLN, and changes in postoperative voice performance.

ELIGIBILITY:
Inclusion Criteria:

* eligible for total thyroidectomy
* no previous history of neck surgery or radiation
* no vocal cord pathology
* no voice disorders

Exclusion Criteria:

* not fit for surgery
* previous history of neck surgery or radiation
* vocal cord pathology
* vocal cord movement disorders

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
rate of identification and exposure of the external laryngeal nerve during thyroidectomy | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No